CLINICAL TRIAL: NCT05220839
Title: Is the Cerclage Area Associated With the Incidence of Preterm Birth in Pregnant Women Undergoing Mc Donald Cerclage?
Brief Title: Relation of the Area of Cerclage With Preterm Birth
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Neval Cayonu, Research fellow in perinatology, Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital
Other Study IDs: 2021/132
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Cervical Insufficiency
Keywords: cerclage area; incidence of preterm birth; Mc Donald
MeSH Terms: conditions — Uterine Cervical Incompetence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Type of cerclage procedure Mc Donald — Patients who underwent Mc Donald cervical cerclage will be calculated the area of cervical cerclage area

SUMMARY:
This study is planned prospectively in pregnancies who applied to Etlik Zübeyde Hanım Women's Health Care, Training and Research Hospital which is a teritiary hospital with 15.000 births anually, between January 2022 and January 2023. Cerclage treatment will be performed with the McDonald technique (the type of cerclage suture will be mersilene) between the 16-23 weeks of gestation in pregnant women with a diagnosis of cervical insufficiency based on the history , physical examination or ultrasound findings according to ACOG. The investigators will measure cerclage area after cerclage treatment (within 0-4 weeks) and different parameters besides it by transvaginal ultrasound. It will be whether the collected data is related to the incidence of preterm birth.

DETAILED DESCRIPTION:
The parameters that will be measured with transvaginal ultrasound are:

* Cerclage area in the axial plane of the cervix
* Angle between anterior uterine wall and internal os
* Angle between anterior uterine wall and external os
* Anterior and posterior cervical widht at level of stitch
* Anterior and posterior stitch depth (stitch to canal )
* Cervical length above and below cerclage stitch

Before the data collection phase ,the required sample number for the research was determined using the G*power (Faul, Erdfelder, Buchner, & Lang, 2009) 3.1 program. When the alpha level is .05 and the power is %95 , the total number of samples was found o be 22.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy between 16-23 weeks of gestation and between the ages of 18-45
* According to ACOG based on history (Having one or more painless abortions between 16-22 weeks of gestation , a history of cerclage
* According to ACOG based on physical examination ( fetal membranes prolapsed from endocervical canal or not, cervical dilation present )
* Accoding to ACOG based on ultrasound examination ( if there is no previous history of preterm birth , if the cervical length is 10mm or less, if the cervical length is less than 25mm with a history of preterm birth )

Exclusion Criteria:

* Multiple pregnancies
* Pregnant women with premature rupture of membranes
* Pregnant women with uterine anomalies
* Pregnant women with fetal anomalies
* Pregnant women with Gestational diabetes mellitus, Chronic or gestational hypertension , fetal growth restriction , oligohydroamnios or polihydroamnios

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients aged between 18-45 years old, have not any maternal chronic ilnesses, have not amnion fluid abnormalities, underwent cervical cerclage according to ACOC criteria between 16-23 gestational weeks.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2023-01-21 (Estimated); Study Completion 2023-02-23 (Estimated)

PRIMARY OUTCOMES:
cervical cerclage area | Between 16-23 weeks of pregnancy
  cervical cerclage will be measured in the axial plane of the cervix by transvaginal ultrasonography
Preterm birth | From date of cervical cerclage to delivery
  The incidence of patients delivered before 37. gestational weeks

CONTACTS AND LOCATIONS:
Overall Officials: Can Tekin Iskender, MD, Study Director — Helath Sciences University, Etlik Zubeyde Hanım Women's Health Training and Research Hospital
Locations (1):
- Etlik Zubeyde Hanım Women's Health Training and Research hospital, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kahraman N, Obut M. Area of cervical cerclage
- See also: my e-mail — http://nevalcayonu@gmail.com